CLINICAL TRIAL: NCT00187187
Title: DAVID II (Dual Chamber and VVI Implantable Defibrillator (DAVID) Trial II)
Acronym: DAVIDII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Heidi Hinrichs, Director of Clinical Operations, St. Jude Medical CRMD
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G990333/SO28
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death; Congestive Heart Failure
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac; Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Implantable Defibrillator (ICD) VVI-40 (Active Comparator): The DAVID II Clinical Study evaluates the hypothesis that, in patients needing an ICD but without overt indications for pacing, AAI pacing with maximal concomitant drug therapy (AAI-70)will not increase the rate of the combined endpoint of mortality or hospitalization for new or worsened heart failure, compared to patients with ventricular backup pacing (VVI-40).
  Interventions: Device: Implantable Defibrillator (ICD)
- Implantable Defibrillator (ICD) AAI-70 (Active Comparator): The DAVID II Clinical Study evaluates the hypothesis that, in patients needing an ICD but without overt indications for pacing, AAI pacing with maximal concomitant drug therapy (AAI-70)will not increase the rate of the combined endpoint of mortality or hospitalization for new or worsened heart failure, compared to patients with ventricular backup pacing (VVI-40).
  Interventions: Device: Implantable Defibrillator (ICD)

INTERVENTIONS:
Device: Implantable Defibrillator (ICD) — Implantable Defibrillator (ICD)
  Other Names: Implantable Defibrillator
  Arms: Implantable Defibrillator (ICD) VVI-40
Device: Implantable Defibrillator (ICD) — Implantable Defibrillator (ICD)
  Arms: Implantable Defibrillator (ICD) AAI-70

SUMMARY:
The DAVID II Clinical Study evaluates the hypothesis that, in patients needing an ICD but without overt indications for pacing, AAI pacing with maximal concomitant drug therapy will not increase the rate of the combined endpoint of mortality or hospitalization for new or worsened heart failure as compared to patients with ventricular backup pacing.

DETAILED DESCRIPTION:
The DAVID II Clinical Study evaluates the hypothesis that, in patients needing an ICD but without overt indications for pacing, AAI pacing with maximal concomitant drug therapy will not increase the rate of the combined endpoint of mortality or hospitalization for new or worsened heart failure, compared to patients with ventricular backup pacing (VVI), and that AAI pacing will result in a reduction of 0.425 years in median event-free survival compared to VVI pacing.

Enrollment and Randomization:

A total of 600 patients have been enrolled and randomized. All patients previously enrolled in the VVI arm of the DAVID Trial who were hemodynamically stable in the VVI-40 programmed mode and willing to participate have been randomized in equal numbers into the study. New patients (not previously randomized in DAVID) have also been enrolled and similarly randomized. The randomization was stratified for investigational site, for previous randomization in DAVID vs being newly-enrolled, for a history of CHF, and, among the new enrollees, for primary versus preventive eligibility criteria.

Patients were enrolled with the same indications used in the DAVID Trial, including MADIT II indications, with the exception that any patient in class III heart failure must have been on optimal heart failure therapy for at least 3 months prior to enrollment and randomization.

Any planned cardiac surgery (ablation, endocardial resection, valve, aneurysmectomy, revascularization) must have been completed before randomization. All patients have received commercially available St. Jude dual chamber ICD systems.

Blinding:

Patients have not be told to which pacing mode, VVI or AAI they have been assigned (i.e., they will be blinded) in order to reduce the potential for patient generated bias in the quality of life assessments which are part of the study.

Crossover:

All patients will remain in the study with the device programmed according to their randomization assignment, from the point of randomization to the end of follow-up. No crossover from one pacing mode to the other is permitted, even after a hospital admission for congestive heart failure, until the reason for the requested crossover is reviewed and permission is obtained from the University of Washington Clinical Trials Center to change pacing mode.

Optimal CHF Pharmacologic Therapy:

Optimal CHF Pharmacologic Therapy in the study consists of digoxin, diuretics, angiotensin-converting enzyme, (ACE) inhibitors , and beta-blockers. Treatment during the study adheres to the Heart Failure Society of America (HFSA) Practice Guidelines. Heart Failure symptoms are treated by adjustment of both the rate and rate response of the pacemaker and the medications.

Primary Endpoint:

The primary endpoint is either death or CHF hospitalization. The determination of CHF hospitalization will be made by an Events Committee based on review of the hospital records blinded as to treatment arm.

Secondary endpoints include:

* Appropriate ICD therapy--ICD shocks plus Antitachycardia Pacing(ATP)events;
* Inappropriate ICD therapy (any therapy deemed not related to Ventricular Tachycardia (VT) or Ventricular Fibrillation (VF);
* Quality of Life (SF-36, MLHF, VAS)

Follow-up:

Patients will be followed at 3-month intervals. The patients are also instructed to call their investigational center any time they receive an ICD shock therapy delivery in order to have an ICD interrogation/download of the device's memory performed.

Data Items Collected:

Standard demographics, clinical histories, and a QoL assessment were obtained at baseline. During the follow-up phase, routine clinical data is obtained every 3 months. Quality of life assessments are be repeated at 6 months. Events (adverse symptoms, hospitalization, death)trigger more extensive data collection including, in particular: 1)all ICD printouts, 2)detailed hospital records for all CHF hospitalizations, and patient records for all deaths.

ELIGIBILITY:
Inclusion Criteria:

I. DAVID I patients enrolled in the VVI-40 who are hemodynamically stable.

II. Patients with an LVEF 0.40 considered for ICD therapy because of one of the following primary, spontaneously occurring, sustained events within the last 6 weeks prior to enrollment:

* VF arrest (ACC/AHA indication Class 1-1),
* VT with syncope (ACC/AHA indication Class 1-1 or 1-2),
* Non-syncopal sustained VT with significant cardiac symptoms or BP < 80 (ACC/AHA indication Class 1-2, IIb-4),

OR

III. Patients considered for ICD therapy because of one of the following:

* LVEF < 0.40 with inducible VT or VF within 6 weeks prior to randomization (with or without spontaneous arrhythmia), or
* LVEF < 0.30 with coronary artery disease, > 1 month from a myocardial infarction, and > 3 months from bypass surgery or percutaneous coronary intervention.

If the ICD was already implanted at time of consideration for enrollment, the device must have been programmed in the VVI mode since implant.

Exclusion Criteria:

* NYHA CHF Class III unless on optimal heart failure therapy for at least 3 months prior to enrollment,
* NYHA CHF Class IV,
* Reversible causes of the VT/VF event,
* Permanent pacemaker,
* First degree AV block with PR interval of more than 240 ms.,
* 2nd or 3rd or advanced degree heart block,
* Symptomatic bradycardia,
* Pre-existing endocardial pacing leads,
* Permanent atrial fibrillation (>= 6 months or unknown duration),
* Patient awaiting a cardiac transplant,
* Life expectancy <1 year,
* Frequent uncontrolled atrial tachyarrhythmia, or
* Inability to obtain informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2003-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is either death or CHF hospitalization. | All 600 enrolled patients will be followed to a common termination date at 2.5 years.
  The primary endpoint is either death or CHF hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Allfred P Hallstrom, PhD, Principal Investigator — University of Washington

REFERENCES:
- [Result] Wilkoff BL, Kudenchuk PJ, Buxton AE, Sharma A, Cook JR, Bhandari AK, Biehl M, Tomassoni G, Leonen A, Klevan LR, Hallstrom AP; DAVID II Investigators. The DAVID (Dual Chamber and VVI Implantable Defibrillator) II trial. J Am Coll Cardiol. 2009 Mar 10;53(10):872-80. doi: 10.1016/j.jacc.2008.10.057. PMID 19264245
- [Result] Kudenchuk PJ, Hallstrom AP, Herre JM, Wilkoff BL; DAVID II Investigators. Heart rate, pacing, and outcome in the Dual Chamber and VVI Implantable Defibrillator (DAVID) trials. Heart Rhythm. 2009 Aug;6(8):1129-35. doi: 10.1016/j.hrthm.2009.04.039. Epub 2009 May 20. PMID 19632624